CLINICAL TRIAL: NCT02537301
Title: Endoscopic Retrograde Cholangiopancreatography(ERCP)-Related Discussion Through a Mobile Social App by Trainees After Finishing ERCP Training
Brief Title: Endoscopic Retrograde Cholangiopancreatography(ERCP)-Related Discussion Through a Mobile Social App by a Group of Doctors
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Other Study IDs: 20150611-4
Record Dates: First submitted 2015-08-13; First posted 2015-09-01 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Endoscopic Retrograde Cholangiopancreatography; social networking; group chat

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ERCP-chat group: All the doctors who finished their ERCP training in Xijing Hospital of Digestive Diseases and were invited to join in a chatting group in a mobile social app (Wechat).
  Interventions: Other: joining in the platform

INTERVENTIONS:
Other: joining in the platform — The activities (contents, chatting frequency etc.) of ERCP doctors on the chatting group were retrospectively extracted. The data related to the performance of ERCP (such as case volume, cannulation success rate and PEP etc.) by ERCP doctors were collected by a questionaire.

SUMMARY:
Group chat through the platform of mobile social networking provides an easily accessible, real-time and interactive channel for communication. With the help of mobile social app, a group of doctors with similar interests can share valuable cases, important papers and opinions through multiple media types (texts, images, and videos). It remains unknown what activities of Endoscopic Retrograde Cholangiopancreatography(ERCP) doctors on a group-chat platform are.

In the beginning of 2013, a chatting group on Wechat (the most popular mobile social app in China), focusing on ERCP, was created. All the doctors who received and finished their ERCP training in Xijing Hospital of Digestive Diseases were invited to join in the platform. The contents in the chatting group were analyzed. The relationships between the chatting activities of ERCP doctors and the performance of ERCP (such as case volume, cannulation success rate and PEP etc.) were investigated.

ELIGIBILITY:
Inclusion Criteria:

* Doctors who received and finished their ERCP training in Xijing Hospital of Digestive Diseases and joined in a chatting group in a mobile social app (Wechat).

Exclusion Criteria:

* Unable to join in the chatting group
* Unable to finish the questionaire
* Denying participating in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Doctors who received and finished their ERCP training in Xijing Hospital of Digestive Diseases and joined in a chatting group through a mobile social app
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Chatting frequency | 1 year

SECONDARY OUTCOMES:
Difficulty grade of the discussed case | 1 year
Number of biliary duct-related cases | 1 year
ERCP performance volumes | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yanglin Pan, Principal Investigator — Xijing Hospital of Disgestive Diseases.The Fourth Military University
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

REFERENCES:
- [Result] Blackmur JP, Clement RG, Brady RR, Oliver CW. Surgical training 2.0: How contemporary developments in information technology can augment surgical training. Surgeon. 2013 Apr;11(2):105-12. doi: 10.1016/j.surge.2012.12.001. Epub 2013 Jan 9. PMID 23312553
- [Result] Ang TL, Cheng J, Khor JL, Mesenas SJ, Vu KF, Wong WK; Endoscopic Retrograde Cholangiopancreatography (ERCP). Guideline on training and credentialing in endoscopic retrograde cholangiopancreatography. Singapore Med J. 2011 Sep;52(9):654-7. PMID 21947141
- [Result] Pan Y, Zhao L, Leung J, Zhang R, Luo H, Wang X, Liu Z, Wan B, Tao Q, Yao S, Hui N, Fan D, Wu K, Guo X. Appropriate time for selective biliary cannulation by trainees during ERCP--a randomized trial. Endoscopy. 2015 Aug;47(8):688-95. doi: 10.1055/s-0034-1391564. Epub 2015 Mar 6. PMID 25750038